CLINICAL TRIAL: NCT04175522
Title: A Phase 2a, Prospective, Open-label, Single-arm, Single Center, Proof of Concept Study to Evaluate the Safety and Efficacy of IGIV 10% in Patients With Autoimmune Encephalitis
Brief Title: Safety and Efficacy of IGIV 10% in Patients With Autoimmune Encephalitis:
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC5107AE01
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Autoimmune Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System | interventions — Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Investigational product(IP)
  Interventions: Drug: Immunoglobulin G

INTERVENTIONS:
Drug: Immunoglobulin G — IGIV 10%(400mg/kg) QD for 5 consecutive days administrated intravenously.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of IGIV 10% in patients with autoimmune encephalitis

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged more than 12 years.(adolescent or adult)
2. Subject who all three of the following diagnosis criteria for possible autoimmune encephalitis have been met.

   * Subacute onset (rapid progression of less than 3 months) of working memory deficits(short-term memory loss), altered mental status, or psychiatric symptoms.
   * At least one of the following:

     * New focal CNS findings
     * Seizure not explained by a previously known seizure disorder
     * CSF pleocytosis (WBC count ≥ 5/mm2)
     * MRI features suggestive of encephalitis
   * Reasonable exclusion of alternative causes
3. Subjects or parent/legal representative willing to provide written informed consent

Exclusion Criteria:

1. Subject who has received Immunoglobulin therapy within 10 weeks prior to screening
2. Subject who has a history of hypersensitivity or shock to ingredient of immunoglobulin
3. Subject who has been diagnosed with IgA deficiency
4. Subject who has renal disorder (creatinine clearance < 10 ml/min) or requires dialysis
5. Subject who has been diagnosed with hemolytic anemia or anemia from blood loss
6. Subject who has been diagnosed with immuonological competence or immunodeficiency
7. Subject who has high risk of thrombus or embolism (History of thrombus/embolism or cerebro/cardiovascular disorder within 3 months prior to screening)
8. Subject who has low heart condition (Congestive heart failure >NYHA functional class Ⅱ: unstable coronary artery disease or myocardiac infarction within 3 months prior to screening)
9. Subject who cannot prohibit the previously administrated steroids by investigator's discretion (ex. Suspicion of steroid dependence, hypoadrenocorticism, when treatment effects are expected, etc.)
10. Females who are pregnant or breast feeding
11. Subject who is considered by investigator to ineligible for the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Chage of mRS(The Modified Rankin Scale) score; 0(better) to 6(worse) | 28 days
  Change of mRS score 7 days and 28 days after IP administration compared with baseline(before IP administration)

SECONDARY OUTCOMES:
Chage and improvement of mRS(The Modified Rankin Scale) score; 0(better) to 6(worse) | 28 days
  Change and improvment of mRS score 14 days and 28 days after IP administration compared with baseline(before IP administration)
Chage and improvement of Glasgow coma scale(GCS); 3(worse) to 15(better) | 28 days
  Change and improvment of Glasgow coma scale(GCS) 7 days, 14 days and 28 days after IP administration compared with baseline(before IP administration)
Chage and improvement of Clinical Global Impression Scale-Severity; 1(better) to 7(worse) | 28 days
  Change and improvment of Clinical Global Impression Scale-Severity 7 days, 14 days and 28 days after IP administration compared with baseline(before IP administration)
Chage and improvement of Clinical Global Impression Scale-Impovement; 1(better) to 7(worse) | 28 days
  Change and improvment of Clinical Global Impression Scale-Improvement 7 days, 14 days and 28 days after IP administration compared with baseline(before IP administration)
Chage and improvement of CASE(Clinical Assessment scale of Encephalitis) score; 0(better) to 27(worse) | 28 days
  Change and improvment of CASE score 7 days, 14 days and 28 days after IP administration compared with baseline(before IP administration)
The relationship | 28 days
  The relationship between neurological scale

CONTACTS AND LOCATIONS:
Overall Officials: Soon Tae Lee, MD, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea